CLINICAL TRIAL: NCT00621855
Title: RandomizEd Dabigatran Etexilate Dose Finding Study in Patients With Acute Coronary Syndromes Post Index Event With Additional Risk Factors for Cardiovascular Complications Also Receiving Aspirin and Clopidogrel: Multi-centre, Prospective, Placebo Controlled, Cohort Dose Escalation Study (RE-DEEM)
Brief Title: RE-DEEM Dose Finding Study for Dabigatran Etexilate in Patients With Acute Coronary Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Uppsala University (Other)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1160.67; RE-DEEM (Other: OTHER); 2007-004301-99 (EudraCT Number: EudraCT)
Record Dates: First submitted 2008-02-13; First posted 2008-02-22 (Estimated); Results first posted 2011-02-11 (Estimated); Last update posted 2014-03-12 (Estimated); Status verified 2014-02

CONDITIONS: Coronary Disease
MeSH Terms: conditions — Coronary Disease | interventions — Dabigatran

ARMS (5):
- Dabigatran etexilate 50mg (Experimental): twice daily dosing,
  Interventions: Drug: dabigatran etexilate
- Dabigatran etexilate 75mg (Experimental): twice daily dosing, patients with moderate renal impairment allocated 50mg bid
  Interventions: Drug: dabigatran etexilate
- Dabigatran etexilate 110mg (Experimental): twice daily dosing, patients with moderate renal impairment allocated 75mg bid
  Interventions: Drug: dabigatran etexilate
- dabigatran etexilate 150mg (Experimental): twice daily dosing, patients with moderate renal impairment allocated 110mg bid
  Interventions: Drug: dabigatran etexilate
- placebo (Placebo Comparator): matched placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: placebo — matched placebo
  Arms: placebo
Drug: dabigatran etexilate — capsules, twice daily, 26 weeks treatment
  Arms: Dabigatran etexilate 50mg
Drug: dabigatran etexilate — capsules, twice daily, 26 weeks treatment
  Arms: Dabigatran etexilate 75mg
Drug: dabigatran etexilate — capsules, twice daily, 26 weeks treatment
  Arms: Dabigatran etexilate 110mg
Drug: dabigatran etexilate — capsules, twice daily, 26 weeks treatment
  Arms: dabigatran etexilate 150mg

SUMMARY:
The purpose of this trial is to evaluate the safety and indicators of efficacy of up to 4 doses of orally administered dabigatran etexilate, administered twice daily, compared to placebo when given in addition to dual antiplatelet treatment in patients with an index event (MI) at high risk for new ischaemic cardiovascular events.

ELIGIBILITY:
Inclusion criteria Patients with acute coronary syndromes with at least one additional risk factor for cardiovascular complications.

Exclusion criteria

1. Long term treatment with any other oral anticoagulant
2. Severe/disabling stroke within last 6 months
3. Conditions associated with increased bleeding risk
4. Anaemia or thrombocytopenia
5. Severe renal impairment
6. Liver disease
7. Positive pregnancy test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1878 (Actual)
Dates: Start 2008-03; Primary Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (167):
- 1160.67.10002 Boehringer Ingelheim Investigational Site, Clearwater, Florida, United States
- Belgium (8):
  - 1160.67.32008 Boehringer Ingelheim Investigational Site, Bouge/Namur
  - 1160.67.32011 Boehringer Ingelheim Investigational Site, Brasschaat
  - 1160.67.32005 Boehringer Ingelheim Investigational Site, Edegem
  - 1160.67.32002 Boehringer Ingelheim Investigational Site, Genk
  - 1160.67.32006 Boehringer Ingelheim Investigational Site, Gilly
  - 1160.67.32003 Boehringer Ingelheim Investigational Site, Hasselt
  - 1160.67.32001 Boehringer Ingelheim Investigational Site, Leuven
  - 1160.67.32004 Boehringer Ingelheim Investigational Site, Tienen
- Bulgaria (11):
  - 1160.67.59007 Boehringer Ingelheim Investigational Site, Burgas
  - 1160.67.59009 Boehringer Ingelheim Investigational Site, Dimitrovgrad
  - 1160.67.59003 Boehringer Ingelheim Investigational Site, Pleven
  - 1160.67.59012 Boehringer Ingelheim Investigational Site, Pleven
  - 1160.67.59006 Boehringer Ingelheim Investigational Site, Rousse
  - 1160.67.59001 Boehringer Ingelheim Investigational Site, Sofia
  - 1160.67.59002 Boehringer Ingelheim Investigational Site, Sofia
  - 1160.67.59004 Boehringer Ingelheim Investigational Site, Sofia
  - 1160.67.59005 Boehringer Ingelheim Investigational Site, Sofia
  - 1160.67.59008 Boehringer Ingelheim Investigational Site, Sofia
  - 1160.67.59010 Boehringer Ingelheim Investigational Site, Sofia
- Canada (12):
  - 1160.67.11009 Boehringer Ingelheim Investigational Site, Calgary, Alberta
  - 1160.67.11003 Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - 1160.67.11012 Boehringer Ingelheim Investigational Site, Cambridge, Ontario
  - 1160.67.11010 Boehringer Ingelheim Investigational Site, Greater Sudbury, Ontario
  - 1160.67.11020 Boehringer Ingelheim Investigational Site, Greater Sudbury, Ontario
  - 1160.67.11008 Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - 1160.67.11018 Boehringer Ingelheim Investigational Site, London, Ontario
  - 1160.67.11017 Boehringer Ingelheim Investigational Site, Mississauga, Ontario
  - 1160.67.11004 Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - 1160.67.11016 Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - 1160.67.11014 Boehringer Ingelheim Investigational Site, Québec, Quebec
  - 1160.67.11006 Boehringer Ingelheim Investigational Site, Terrebonne, Quebec
- Czechia (6):
  - 1160.67.42007 Boehringer Ingelheim Investigational Site, Hradec Králové
  - 1160.67.42005 Boehringer Ingelheim Investigational Site, Litoměřice
  - 1160.67.42008 Boehringer Ingelheim Investigational Site, Ostrava
  - 1160.67.42001 Boehringer Ingelheim Investigational Site, Prague
  - 1160.67.42003 Boehringer Ingelheim Investigational Site, Teplice
  - 1160.67.42002 Boehringer Ingelheim Investigational Site, Zlín
- Denmark (4):
  - 1160.67.45001 Boehringer Ingelheim Investigational Site, Aarhus C
  - 1160.67.45003 Boehringer Ingelheim Investigational Site, Hvidovre
  - 1160.67.45002 Boehringer Ingelheim Investigational Site, Odense
  - 1160.67.45004 Boehringer Ingelheim Investigational Site, Roskilde
- Finland (4):
  - 1160.67.58001 Boehringer Ingelheim Investigational Site, HUS
  - 1160.67.58004 Boehringer Ingelheim Investigational Site, Jyväskylä
  - 1160.67.58003 Boehringer Ingelheim Investigational Site, Kuopio
  - 1160.67.58002 Boehringer Ingelheim Investigational Site, Pori
- France (7):
  - 1160.67.3305A Boehringer Ingelheim Investigational Site, Brest
  - 1160.67.3305B Boehringer Ingelheim Investigational Site, Brest
  - 1160.67.3303A Boehringer Ingelheim Investigational Site, Dijon
  - 1160.67.3303B Boehringer Ingelheim Investigational Site, Dijon
  - 1160.67.3303C Boehringer Ingelheim Investigational Site, Dijon
  - 1160.67.3303D Boehringer Ingelheim Investigational Site, Dijon
  - 1160.67.3301A Boehringer Ingelheim Investigational Site, Paris
- Georgia (6):
  - 1160.67.95001 Boehringer Ingelheim Investigational Site, Tbilisi
  - 1160.67.95002 Boehringer Ingelheim Investigational Site, Tbilisi
  - 1160.67.95003 Boehringer Ingelheim Investigational Site, Tbilisi
  - 1160.67.95004 Boehringer Ingelheim Investigational Site, Tbilisi
  - 1160.67.95005 Boehringer Ingelheim Investigational Site, Tbilisi
  - 1160.67.95006 Boehringer Ingelheim Investigational Site, Tbilisi
- Germany (8):
  - 1160.67.49001 Boehringer Ingelheim Investigational Site, Berlin
  - 1160.67.49007 Boehringer Ingelheim Investigational Site, Berlin
  - 1160.67.49017 Boehringer Ingelheim Investigational Site, Dresden
  - 1160.67.49006 Boehringer Ingelheim Investigational Site, Hanover
  - 1160.67.49019 Boehringer Ingelheim Investigational Site, Homburg/Saar
  - 1160.67.49008 Boehringer Ingelheim Investigational Site, Ludwigshafen am Rhein
  - 1160.67.49015 Boehringer Ingelheim Investigational Site, Neuss
  - 1160.67.49004 Boehringer Ingelheim Investigational Site, Rostock
- Hungary (9):
  - 1160.67.36001 Boehringer Ingelheim Investigational Site, Budapest
  - 1160.67.36003 Boehringer Ingelheim Investigational Site, Budapest
  - 1160.67.36004 Boehringer Ingelheim Investigational Site, Budapest
  - 1160.67.36002 Boehringer Ingelheim Investigational Site, Debrecen
  - 1160.67.36007 Boehringer Ingelheim Investigational Site, Kecskemét
  - 1160.67.36006 Boehringer Ingelheim Investigational Site, Komárom
  - 1160.67.36008 Boehringer Ingelheim Investigational Site, Miskolc
  - 1160.67.36009 Boehringer Ingelheim Investigational Site, Mosonmagyaróvár
  - 1160.67.36005 Boehringer Ingelheim Investigational Site, Zalaegerszeg
- India (7):
  - 1160.67.91004 Boehringer Ingelheim Investigational Site, Amedabad
  - 1160.67.91001 Boehringer Ingelheim Investigational Site, Chennai
  - 1160.67.91005 Boehringer Ingelheim Investigational Site, Hyderabad
  - 1160.67.91007 Boehringer Ingelheim Investigational Site, Lucknow
  - 1160.67.91002 Boehringer Ingelheim Investigational Site, Mumbai
  - 1160.67.91003 Boehringer Ingelheim Investigational Site, Pune
  - 1160.67.91006 Boehringer Ingelheim Investigational Site, Pune
- Ireland (2):
  - 1160.67.53001 Boehringer Ingelheim Investigational Site, Dublin
  - 1160.67.53002 Boehringer Ingelheim Investigational Site, Dublin
- Italy (6):
  - 1160.67.39006 Boehringer Ingelheim Investigational Site, Ascoli Piceno
  - 1160.67.39003 Boehringer Ingelheim Investigational Site, Milan
  - 1160.67.39005 Boehringer Ingelheim Investigational Site, Milan
  - 1160.67.39001 Boehringer Ingelheim Investigational Site, Parma
  - 1160.67.39002 Boehringer Ingelheim Investigational Site, S. Maria Capua Vetere (CE)
  - 1160.67.39004 Boehringer Ingelheim Investigational Site, Torino
- Netherlands (10):
  - 1160.67.31003 Boehringer Ingelheim Investigational Site, 's-Hertogenbosch
  - 1160.67.31001 Boehringer Ingelheim Investigational Site, Amsterdam
  - 1160.67.31009 Boehringer Ingelheim Investigational Site, Ede
  - 1160.67.31002 Boehringer Ingelheim Investigational Site, Groningen
  - 1160.67.31006 Boehringer Ingelheim Investigational Site, Helmond
  - 1160.67.31011 Boehringer Ingelheim Investigational Site, Hoogeveen
  - 1160.67.31005 Boehringer Ingelheim Investigational Site, Rotterdam
  - 1160.67.31008 Boehringer Ingelheim Investigational Site, Spijkenisse
  - 1160.67.31007 Boehringer Ingelheim Investigational Site, The Hague
  - 1160.67.31004 Boehringer Ingelheim Investigational Site, Tilburg
- Norway (5):
  - 1160.67.47005 Boehringer Ingelheim Investigational Site, Drammen
  - 1160.67.47002 Boehringer Ingelheim Investigational Site, Hamar
  - 1160.67.47003 Boehringer Ingelheim Investigational Site, Haugesund
  - 1160.67.47004 Boehringer Ingelheim Investigational Site, Hønefoss
  - 1160.67.47001 Boehringer Ingelheim Investigational Site, Oslo
- Poland (6):
  - 1160.67.48003 Boehringer Ingelheim Investigational Site, Bydgoszcz
  - 1160.67.48006 Boehringer Ingelheim Investigational Site, Bydgoszcz
  - 1160.67.48004 Boehringer Ingelheim Investigational Site, Gdynia
  - 1160.67.48005 Boehringer Ingelheim Investigational Site, Inowrocław
  - 1160.67.48002 Boehringer Ingelheim Investigational Site, Sopot
  - 1160.67.48001 Boehringer Ingelheim Investigational Site, Warsaw
- Romania (7):
  - 1160.67.40006 Boehringer Ingelheim Investigational Site, Baia Mare
  - 1160.67.40005 Boehringer Ingelheim Investigational Site, Brăila
  - 1160.67.40001 Boehringer Ingelheim Investigational Site, Bucharest
  - 1160.67.40003 Boehringer Ingelheim Investigational Site, Bucharest
  - 1160.67.40004 Boehringer Ingelheim Investigational Site, Bucharest
  - 1160.67.40002 Boehringer Ingelheim Investigational Site, Oradea
  - 1160.67.40007 Boehringer Ingelheim Investigational Site, Tg. Mures
- Russia (11):
  - 1160.67.70001 Boehringer Ingelheim Investigational Site, Moscow
  - 1160.67.70002 Boehringer Ingelheim Investigational Site, Moscow
  - 1160.67.70003 Boehringer Ingelheim Investigational Site, Moscow
  - 1160.67.70004 Boehringer Ingelheim Investigational Site, Moscow
  - 1160.67.70005 Boehringer Ingelheim Investigational Site, Moscow
  - 1160.67.70006 Boehringer Ingelheim Investigational Site, Moscow
  - 1160.67.70007 Boehringer Ingelheim Investigational Site, Moscow
  - 1160.67.70008 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1160.67.70009 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1160.67.70010 Boehringer Ingelheim Investigational Site, Saratov
  - 1160.67.70011 Boehringer Ingelheim Investigational Site, Saratov
- South Korea (13):
  - 1160.67.82010 Boehringer Ingelheim Investigational Site, Busan
  - 1160.67.82008 Boehringer Ingelheim Investigational Site, Daegu
  - 1160.67.82009 Boehringer Ingelheim Investigational Site, Daegu
  - 1160.67.82013 Boehringer Ingelheim Investigational Site, Daejeon
  - 1160.67.82006 Boehringer Ingelheim Investigational Site, Daejoen
  - 1160.67.82007 Boehringer Ingelheim Investigational Site, Incheon
  - 1160.67.82012 Boehringer Ingelheim Investigational Site, Jeonju
  - 1160.67.82005 Boehringer Ingelheim Investigational Site, Kwangju
  - 1160.67.82011 Boehringer Ingelheim Investigational Site, Pusan
  - 1160.67.82001 Boehringer Ingelheim Investigational Site, Seoul
  - 1160.67.82002 Boehringer Ingelheim Investigational Site, Seoul
  - 1160.67.82003 Boehringer Ingelheim Investigational Site, Seoul
  - 1160.67.82004 Boehringer Ingelheim Investigational Site, Seoul
- Spain (6):
  - 1160.67.34001 Boehringer Ingelheim Investigational Site, Barcelona
  - 1160.67.34002 Boehringer Ingelheim Investigational Site, Barcelona
  - 1160.67.34005 Boehringer Ingelheim Investigational Site, Madrid
  - 1160.67.34006 Boehringer Ingelheim Investigational Site, Madrid
  - 1160.67.34003 Boehringer Ingelheim Investigational Site, Sabadell (Barcelona)
  - 1160.67.34004 Boehringer Ingelheim Investigational Site, Tarragona
- Sweden (7):
  - 1160.67.46004 Boehringer Ingelheim Investigational Site, Gothenburg
  - 1160.67.46006 Boehringer Ingelheim Investigational Site, Gothenburg
  - 1160.67.46007 Boehringer Ingelheim Investigational Site, Malmo
  - 1160.67.46005 Boehringer Ingelheim Investigational Site, Motala
  - 1160.67.46002 Boehringer Ingelheim Investigational Site, Stockholm
  - 1160.67.46001 Boehringer Ingelheim Investigational Site, Uppsala
  - 1160.67.46003 Boehringer Ingelheim Investigational Site, Vaesteraas
- Ukraine (8):
  - 1160.67.38002 Boehringer Ingelheim Investigational Site, Ivano-Frankivsk
  - 1160.67.38004 Boehringer Ingelheim Investigational Site, Kharkiv
  - 1160.67.38007 Boehringer Ingelheim Investigational Site, Kharkiv
  - 1160.67.38001 Boehringer Ingelheim Investigational Site, Kiev
  - 1160.67.38003 Boehringer Ingelheim Investigational Site, Kiev
  - 1160.67.38005 Boehringer Ingelheim Investigational Site, Kiev
  - 1160.67.38008 Boehringer Ingelheim Investigational Site, Nikolayev
  - 1160.67.38006 Boehringer Ingelheim Investigational Site, Odesa
- United Kingdom (3):
  - 1160.67.44003 Boehringer Ingelheim Investigational Site, Brighton
  - 1160.67.44002 Boehringer Ingelheim Investigational Site, Exeter
  - 1160.67.44001 Boehringer Ingelheim Investigational Site, Middlesbrough

RESULTS

PARTICIPANT FLOW:
Recruitment Details: International multi-centre trial with 161 trial sites in 24 countries recruiting patients with acute coronary syndromes with increased troponin levels within 14 days post index myocardial infarction (ST or non-ST elevation between March 2008 and March 2009.
Pre-assignment Details: Patients receiving aspirin and clopidogrel at randomisation were included. They also had at least 1 additional risk factor (for e.g. age ≥65 years, diabetes previous myocardial infarction, peripheral arterial disease). Moderate renal impairment at screening resulted in dose adjustment.
Groups:
- 50mg Dabigatran Etexilate; 75mg Dabigatran Etexilate; 110mg Dabigatran Etexilate; 150mg Dabigatran Etexilate; Placebo: 26 week blinded treatment
Period: Overall Study
Arm/Group | 50mg Dabigatran Etexilate | 75mg Dabigatran Etexilate | 110mg Dabigatran Etexilate | 150mg Dabigatran Etexilate | Placebo
Started | 372 (Started means randomised to treatment) | 371 (Started means randomised to treatment) | 411 (Started means randomised to treatment) | 351 (Started means randomised to treatment) | 373 (Started means randomised to treatment)
Completed | 296 (Completed means completed treatment) | 310 (Completed means completed treatment) | 330 (Completed means completed treatment) | 284 (Completed means completed treatment) | 318 (Completed means completed treatment)
Not Completed | 76 | 61 | 81 | 67 | 55
Not completed — Adverse Event | 32 | 31 | 48 | 34 | 31
Not completed — Lost to Follow-up | 0 | 1 | 3 | 4 | 1
Not completed — Protocol Violation | 16 | 8 | 6 | 7 | 8
Not completed — Withdrawal by Subject | 16 | 11 | 13 | 13 | 9
Not completed — Other | 9 | 7 | 6 | 5 | 4
Not completed — Patients did not receive study drug | 3 | 3 | 5 | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 50mg Dabigatran Etexilate | 75mg Dabigatran Etexilate | 110mg Dabigatran Etexilate | 150mg Dabigatran Etexilate | Placebo | Total
Number analyzed (Participants) | 372 | 371 | 411 | 351 | 373 | 1878
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.9 (12.2) | 60.7 (11.7) | 62.3 (11.1) | 62.3 (10.8) | 61.5 (11.3) | 61.8 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 75 | 117 | 93 | 81 | 450
  Male | 288 | 296 | 294 | 258 | 292 | 1428
Race (NIH/OMB) [Number; unit: participants]
  White | 288 | 267 | 324 | 300 | 268 | 1447
  Black | 0 | 1 | 0 | 0 | 0 | 1
  Asian | 84 | 102 | 82 | 51 | 105 | 424
  Other | 0 | 1 | 5 | 0 | 0 | 6
Region of Enrollment [Number; unit: participants]
  Central Europe | 165 | 155 | 230 | 217 | 165 | 932
  Western Europe | 98 | 93 | 79 | 72 | 84 | 426
  Asia | 84 | 99 | 81 | 51 | 104 | 419
  North America | 25 | 24 | 21 | 11 | 20 | 101
Type of Index Event [Number; unit: participants]
  ST elevation myocardial infarction (STEMI) | 211 | 227 | 254 | 204 | 230 | 1126
  Non ST elevation myocardial infarction (NSTEMI) | 161 | 144 | 157 | 147 | 143 | 752
Creatinine Clearance N=(372;371;411;350;373;1877) [Mean (Standard Deviation); unit: mL/min] | 85.4 (30.2) | 88.7 (32.4) | 84.7 (32) | 86.3 (28.1) | 86.6 (34.8) | 86.3 (31.6)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Displaying the Composite of Major and Clinically Relevant Minor Bleeding Events During Total Observation Time
Description: International Society Thrombosis and Haemostasis (ISTH) definition of a major bleed, and clinically relevant minor bleed.
  A bleeding event was considered as major if it was fatal, was a symptomatic bleeding in a critical area or organ (intracranial, intraspinal, intraocular, retroperitoneal, intra-articular, pericardial, or intramuscular with compartment syndrome), or caused a fall in haemoglobin level of ≥2 g/dL (≥1.24 mmol/L), or led to transfusion of ≥2 units of whole blood or red cells.
  All non major bleeding events were classified as minor bleeds; minor bleeds were subdivided in clinically relevant minor bleeds and not clinically relevant minor bleeds. A CRBE was defined as an acute or subacute clinically overt bleed that did not meet the criteria of a major bleed but either lead to hospital admission and/or a physician guided medical or surgical treatment and/or a change in antithrombotic therapy (including interruption or discontinuation of study drug).
Time Frame: 6 month treatment period + 2 week post treatment follow up
Population: Treated set - The treated set includes all patients who received at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | 50mg Dabigatran Etexilate | 75mg Dabigatran Etexilate | 110mg Dabigatran Etexilate | 150mg Dabigatran Etexilate | Placebo
Number analyzed (Participants) | 369 | 368 | 406 | 347 | 371
participants
  Major and clinically relevant minor bleed events | 13 | 16 | 32 | 27 | 8
  No major or clinically relevant minor bleed events | 356 | 352 | 374 | 320 | 363
Statistical Analysis 1: Comparison: 50mg Dabigatran Etexilate vs 75mg Dabigatran Etexilate vs 110mg Dabigatran Etexilate vs 150mg Dabigatran Etexilate vs Placebo; The proportion of patients who reach this endpoint were analysed by a logistic model for linear trend (dose response). The null hypothesis is that the relationship between dose level (0mg, 50mg, 75mg, 110mg and 150mg) and the proportions of patients with major and clinically relevant minor bleeding is not linear (slope parameter = 0); Test type: Superiority or Other; p < 0.001, Cochran-Armitage test for linear trend

2. Secondary Outcome: Composite of Cardiovascular Death (CVD) With Non Fatal Myocardial Infarction (MI) and Non Haemorrhagic Stroke and All Cause Death (ACD), Non Fatal MI, Severe Recurrent Ischaemia (SRI) and Non Haemorrhagic Stroke During Six Months Treatment
Description: Number of Participants with Composite of Cardiovascular death (CVD) with non fatal myocardial infarction (MI) and non haemorrhagic stroke and All cause death (ACD), non fatal MI, severe recurrent ischaemia (SRI) and non haemorrhagic stroke during six months treatment
Time Frame: 6 month treatment period + 2 week post treatment follow up
Population: Treated set
Measure: Number; unit: participants
Arm/Group | 50mg Dabigatran Etexilate | 75mg Dabigatran Etexilate | 110mg Dabigatran Etexilate | 150mg Dabigatran Etexilate | Placebo
Number analyzed (Participants) | 369 | 368 | 406 | 347 | 371
participants
  CVD, non-fatal MI, non-haemorrhagic stroke | 17 | 18 | 12 | 12 | 14
  ACD, non-fatal MI, SRI, non-haemorrhagic stroke | 25 | 27 | 21 | 25 | 26

3. Secondary Outcome: Individual Occurrence of Death (Cardiovascular and All-cause), Non-fatal MI, Severe Recurrent Ischaemia and Non-haemorrhagic Stroke During Six Months of Treatment
Description: Number of Participants with individual occurrence of death (cardiovascular and all-cause), non-fatal MI, severe recurrent ischaemia and non-haemorrhagic stroke during six months of treatment.
Time Frame: 6 month treatment period + 2 week post treatment follow up
Population: Treated set
Measure: Number; unit: participants
Arm/Group | 50mg Dabigatran Etexilate | 75mg Dabigatran Etexilate | 110mg Dabigatran Etexilate | 150mg Dabigatran Etexilate | Placebo
Number analyzed (Participants) | 369 | 368 | 406 | 347 | 371
participants
  Cardiovascular death | 8 | 9 | 5 | 4 | 9
  Non-fatal myocardial infarction | 9 | 8 | 7 | 8 | 4
  Severe recurrent ischaemia | 9 | 11 | 9 | 11 | 9
  Non-haemorrhagic stroke | 0 | 1 | 0 | 0 | 3
  All cause death | 8 | 10 | 7 | 7 | 14

4. Secondary Outcome: Number of Participants With Any Reduction of D-dimer Concentration
Time Frame: at 1 week and 4 weeks
Population: Full analysis set - The full analysis set includes all randomised and treated patients who had at least one post-dose assessment of D-dimer available.
Measure: Number; unit: participants
Arm/Group | 50mg Dabigatran Etexilate | 75mg Dabigatran Etexilate | 110mg Dabigatran Etexilate | 150mg Dabigatran Etexilate | Placebo
Number analyzed (Participants) | 358 | 358 | 388 | 332 | 356
participants
  Number of Patients with any reduction | 290 | 293 | 333 | 296 | 264
  Number of Patients with no reduction | 48 | 49 | 41 | 28 | 77
  Missing data | 20 | 16 | 14 | 8 | 15
Statistical Analysis 1: Comparison: 50mg Dabigatran Etexilate vs 75mg Dabigatran Etexilate vs 110mg Dabigatran Etexilate vs 150mg Dabigatran Etexilate vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Cochran-Armitage test for linear trend

5. Secondary Outcome: Change From Baseline in log10 D-dimer After 1 and 4 Weeks
Description: Change from baseline in log10 D-dimer concentration after 1 and 4 weeks of dabigatran etexilate treatment compared to placebo. The standard deviation is the geometric standard deviation.
Time Frame: Baseline and at 1 week and 4 weeks
Population: Full Analysis Set (FAS)
Measure: Geometric Mean (Standard Deviation); unit: ratio
Arm/Group | 50mg Dabigatran Etexilate | 75mg Dabigatran Etexilate | 110mg Dabigatran Etexilate | 150mg Dabigatran Etexilate | Placebo
Number analyzed (Participants) | 358 | 358 | 388 | 332 | 356
ratio
  Ratio of week 4 to baseline | 0.33 (3.04) | 0.31 (3.30) | 0.29 (3.14) | 0.31 (3.02) | 0.57 (3.01)
  Ratio of week 1 to baseline | 0.58 (2.60) | 0.52 (2.81) | 0.52 (2.54) | 0.55 (2.58) | 0.87 (2.45)

6. Secondary Outcome: Number of Participants With Bleeding Events During Total Observation Time
Description: International Society Thrombosis and Haemostasis (ISTH) definition of a major bleed, and clinically relevant minor bleed.
  A bleeding event was considered as major if it was fatal, was a symptomatic bleeding in a critical area or organ (intracranial, intraspinal, intraocular, retroperitoneal, intra-articular, pericardial, or intramuscular with compartment syndrome), or caused a fall in haemoglobin level of ≥2 g/dL (≥1.24 mmol/L), or led to transfusion of ≥2 units of whole blood or red cells.
  All non major bleeding events were classified as minor bleeds; minor bleeds were subdivided in clinically relevant minor bleeds (CRBE) and not clinically relevant minor bleeds. A CRBE was defined as an acute or subacute clinically overt bleed that did not meet the criteria of a major bleed but either lead to hospital admission and/or a physician guided medical or surgical treatment and/or a change in antithrombotic therapy (including interruption or discontinuation of study drug).
Time Frame: 6 month treatment period + 2 week post treatment follow up
Population: Treated set
Measure: Number; unit: participants
Arm/Group | 50mg Dabigatran Etexilate | 75mg Dabigatran Etexilate | 110mg Dabigatran Etexilate | 150mg Dabigatran Etexilate | Placebo
Number analyzed (Participants) | 369 | 368 | 406 | 347 | 371
participants
  Major bleeding events | 3 | 1 | 8 | 4 | 2
  Clinically relevant bleeding events | 10 | 16 | 24 | 23 | 6
  Not clinically relevant bleeding events | 32 | 29 | 35 | 20 | 17
  Any bleeding events | 42 | 45 | 60 | 42 | 25

7. Secondary Outcome: Laboratory Analyses
Description: Number of patients with possible clinically significant abnormalities. Clinically significant abnormalities refers to the increase or decrease from baseline.
Time Frame: 6 month treatment period + 2 week post treatment follow up
Population: Treated set
Measure: Number; unit: participants
Arm/Group | 50mg Dabigatran Etexilate | 75mg Dabigatran Etexilate | 110mg Dabigatran Etexilate | 150mg Dabigatran Etexilate | Placebo
Number analyzed (Participants) | 369 | 368 | 406 | 347 | 371
participants
  AST increase N=(359;359;388;329;356) | 8 | 5 | 5 | 2 | 4
  AST decrease N=(359;359;388;329;356) | 0 | 0 | 0 | 0 | 0
  ALT increase N=(359;359;388;329;356) | 10 | 4 | 4 | 7 | 4
  ALT decrease N=(359;359;388;329;356) | 0 | 0 | 0 | 0 | 0
  Bilirubin increase N=(359;360;388;329;355) | 1 | 1 | 2 | 0 | 0
  Bilirubin decrease N=(359;360;388;329;355) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 month treatment period + 3 days
Arm/Group | 50mg Dabigatran Etexilate | 75mg Dabigatran Etexilate | 110mg Dabigatran Etexilate | 150mg Dabigatran Etexilate | Placebo
Serious Adverse Events (participants affected / at risk) | 33/369 | 31/368 | 35/406 | 21/347 | 32/371
Other Adverse Events (participants affected / at risk) | 0/369 | 0/368 | 0/406 | 0/347 | 0/371
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 50mg Dabigatran Etexilate (N=369) | 75mg Dabigatran Etexilate (N=368) | 110mg Dabigatran Etexilate (N=406) | 150mg Dabigatran Etexilate (N=347) | Placebo (N=371)
angina pectoris (Cardiac disorders) | 1 (1) | 4 (5) | 3 (3) | 2 (2) | 5 (5)
Unstable angina (Cardiac disorders) | 4 (4) | 4 (4) | 2 (2) | 1 (1) | 1 (1)
cardiac failure (Cardiac disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
acute cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
coronary artery stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
acute LV failure (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
1st degree AV block (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
congestive cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
cardiac tamponade (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
coronary artery disease (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
coronary artery occlusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
coronary artery thrombosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LV failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
post infarct angina (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ventricular fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Coronary artery insufficiency (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
chest pain (General disorders) | 3 (3) | 4 (5) | 1 (1) | 0 (0) | 1 (1)
non cardiac chest pain (General disorders) | 1 (1) | 1 (1) | 3 (3) | 2 (2) | 1 (1)
asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
bacterial arthritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
infective cholecystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
diabetic gangrene (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
diverticuliitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
lobar pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ischaemia (Vascular disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
angiopathy (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BP fluctuation (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
extremity necrosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
peripheral ischaemia (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
reflux oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
erosive gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
acute cholecystitis (Hepatobiliary disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
bile duct stone (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
hydrocholecystis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
acetabulum fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
in stent coronary artery stenosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
lead dislodgement (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
inadequate control of diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
hemianopia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
paraparesis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
acute prerenal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
acute renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
thrombocythaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
haemoglobin decrease (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.